CLINICAL TRIAL: NCT04023994
Title: A Single-Center, Randomized, Adaptive, Investigator/Subject Blind, Single Ascending Dose, Placebo-Controlled Phase I Study to Investigate the Safety, Tolerability, Immunogenicity and Pharmacokinetics of Intravenously Administered RO7126209 in Healthy Participants
Brief Title: A Single Ascending Dose Study to Investigate the Safety, Tolerability, Immunogenicity and Pharmacokinetics of Intravenously Administered RO7126209 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP41192
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): In Cohorts 1-5, there were ten participants in total who received placebo, two in each cohort.
  Interventions: Drug: Placebo
- RO7126209 (0.1 mg/kg) (Experimental): Healthy volunteers will be administered a single intravenous dose of RO7126209 (0.1 mg/kg).
  Interventions: Drug: RO7126209
- RO7126209 (0.4 mg/kg) (Experimental): Healthy volunteers will be administered a single intravenous dose of RO7126209 (0.4 mg/kg).
  Interventions: Drug: RO7126209
- RO7126209 (1.2 mg/kg) (Experimental): Healthy volunteers will be administered a single intravenous dose of RO7126209 (1.2 mg/kg).
  Interventions: Drug: RO7126209
- RO7126209 (3.6 mg/kg) (Experimental): Healthy volunteers will be administered a single intravenous dose of RO7126209 (3.6 mg/kg).
  Interventions: Drug: RO7126209
- RO7126209 (7.2 mg/kg) (Experimental): Healthy volunteers will be administered a single intravenous dose of RO7126209 (7.2 mg/kg).
  Interventions: Drug: RO7126209

INTERVENTIONS:
Drug: RO7126209 — Participants will be administered single-ascending intravenous doses of RO7126209 with at least 2 weeks between each dose level. After the starting dose, the subsequent doses will be selected in an adaptive design. Sentinel dosing will be employed.
  Arms: RO7126209 (0.1 mg/kg); RO7126209 (0.4 mg/kg); RO7126209 (1.2 mg/kg); RO7126209 (3.6 mg/kg); RO7126209 (7.2 mg/kg)
Drug: Placebo — Participants will be administered a single intravenous dose of matching placebo.
  Arms: Placebo

SUMMARY:
Study BP41192 is a randomized, adaptive, placebo-controlled parallel group study to investigate the safety, tolerability, immunogenicity and pharmacokinetics of single-ascending intravenous (IV) doses of RO7126209 in healthy participants. RO7126209 is being developed for the treatment of Alzheimer's Disease.

DETAILED DESCRIPTION:
This study uses a parallel group design, with participants recruited in 5 planned sequential cohorts. Additional cohort(s) may be added if dose escalation stopping criteria are not met after cohort 5. Participants will receive a single IV dose of either RO7126209 or placebo. RO7126209 doses will be administered in ascending order. After the starting dose, subsequent doses will be selected in an adaptive manner during study conduct based on emerging safety, tolerability and PK data.

ELIGIBILITY:
Inclusion Criteria:

* Healthy status is defined by the absence of evidence of any active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, ophthalmologic examination, hematology, blood chemistry, coagulation, serology, and urinalysis.
* Body mass index (BMI) of 18-30 kg/m2 inclusive
* During the treatment period and until the final follow up visit, agreement to: (1) Remain abstinent or use contraceptive measures such as a condom plus an additional contraceptive method that together result in a failure rate of <1% per year, with a partner who is a woman of childbearing potential. (2) With pregnant female partner, remain abstinent or use contraceptive measures such as a condom to avoid exposing the embryo. (3) Refrain from donating sperm from Day 1 of the study until 90 days after last dose.

Exclusion Criteria:

* Concomitant disease or condition that could interfere with, or treatment of which might interfere with, the conduct of the study, or that would, in the opinion of the Investigator, pose an unacceptable risk to the participant in this study.
* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, ophthalmologic, hematological or allergic disease, metabolic disorder, cancer or cirrhosis.
* Any suspicion or history of alcohol abuse and/or suspicion of regular consumption of drug of abuse within the last 5 years.
* Positive result on hepatitis B (HBV), hepatitis C (HCV), or human immunodeficiency virus (HIV) 1 and 2.
* History or presence of clinically significant ECG abnormalities or cardiovascular disease.
* Clinically-significant abnormalities in laboratory test results.
* Any major illness within one month before the screening examination or any febrile illness within one week prior to screening and up to first dose administration.
* Impaired hepatic function as indicated by screening aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >=1.5 x the upper limit of normal (ULN) or abnormal total bilirubin unless due to Gilbert's disease.
* Any clinically relevant history of hypersensitivity or allergic reactions, either spontaneous or following drug administration, or exposure to foods or environmental agents.
* History of hypersensitivity to biologic agents or any of the excipients in the formulation.
* History of raised intra-cerebral pressure or vertebral joint pathology
* Use of prohibited medication or herbal remedies as described in the section of concomitant medications
* Prior administration of gantenerumab (RO4909832)
* Any vaccination within two months prior to Day 1
* Participation in an investigational drug medicinal product or medical device study within 30 days before screening or within seven times the elimination half-life if known, whichever is longer.
* Participants who regularly smoke more than 5 cigarettes daily or equivalent and are unable or unwilling not to smoke during the in-house period.
* Donation or loss of blood over 500 mL within three months prior to Day 1 and donation of blood for the duration of the study until follow-up.
* Evidence of clinically significant brain magnetic resonance imaging (MRI) findings, including lacunar infarct, territorial infarct or macroscopic hemorrhage, microbleed or area of leptomeningeal hemosiderosis, or deep white matter lesions corresponding to an overall Fazekas score of ≥ 2.
* Claustrophobia, presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body that would contraindicate an MRI scan.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-08-03 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- PRA Health Sciences, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 center in 1 country.
Pre-assignment Details: A total of 36 participants were enrolled at 1 site in the US, out of which 26 participants received active treatment while 10 received placebo.
Groups:
- RO7126209 (0.1 mg/kg): Healthy volunteers were administered a single intravenous dose of RO7126209 (0.1 mg/kg).
- RO7126209 (0.4 mg/kg): Healthy volunteers were administered a single intravenous dose of RO7126209 (0.4 mg/kg).
- RO7126209 (1.2 mg/kg): Healthy volunteers were administered a single intravenous dose of RO7126209 (1.2 mg/kg).
- RO7126209 (3.6 mg/kg): Healthy volunteers were administered a single intravenous dose of RO7126209 (3.6 mg/kg).
- RO7126209 (7.2 mg/kg): Healthy volunteers were administered a single intravenous dose of RO7126209 (7.2 mg/kg).
Period: Overall Study
Arm/Group | Placebo | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Started | 10 | 4 | 4 | 6 | 6 | 6
Completed | 10 | 3 | 2 | 5 | 6 | 6
Not Completed | 0 | 1 | 2 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg) | Total
Number analyzed (Participants) | 10 | 4 | 4 | 6 | 6 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (6.6) | 30.8 (5.9) | 23.5 (4.5) | 24.2 (3.8) | 33.0 (5.9) | 33.3 (2.6) | 29.2 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 4 | 4 | 6 | 6 | 6 | 36
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnicity
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 3
    Not Hispanic or Latino | 10 | 4 | 4 | 6 | 5 | 4 | 33
Race/Ethnicity, Customized [Number; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Asian | 2 | 0 | 0 | 0 | 1 | 0 | 3
    Black or African American | 3 | 1 | 3 | 3 | 2 | 1 | 13
    White | 5 | 2 | 1 | 1 | 3 | 4 | 16
    Multiple | 0 | 1 | 0 | 1 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An Adverse Event can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as Adverse Events.
Time Frame: Up to approximately 9 weeks
Population: The Safety Population was defined as all participants randomised to study treatment and who received at least one dose of the study treatment, whether prematurely withdrawn from the study or not.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 10 | 4 | 4 | 6 | 6 | 6
Percentage of Participants | 80.0 | 75.0 | 50.0 | 83.3 | 100.0 | 100.0

2. Secondary Outcome: Concentration at the End of Infusion (Cend) of RO7126209
Description: Plasma concentrations of RO7126209 were measured by a specific and validated assay at specified timepoints. Plasma PK parameters of RO7126209 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods. Geometric Mean and Coefficient of Variation data are presented below.
Time Frame: Day 1
Population: The PK Analysis population was defined as all participants who received active (RO7126209) treatment. Participants were excluded from the PK analysis population if they significantly violated the inclusion or exclusion criteria, deviated significantly from the protocol, or if data were unavailable or incomplete which could have influenced the PK analysis. Data presented below is only for participants included in the actual analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
µg/mL | 1.80 (15.9) | 7.93 (21.3) | 22.2 (17.6) | 85.7 (22.9) | 160 (26.5)

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 h Postdose (AUC0-24h) of RO7126209
Description: Plasma concentrations of RO7126209 were measured by a specific and validated assay. Plasma PK parameters of RO7126209 were read directly from the plasma concentration versus time profiles or calculated by using standard non-compartmental methods. Geometric Mean and Coefficient of Variation data are presented below.
Time Frame: Days 1 and 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
hr.µg/mL | 27.1 (23.2) | 124 (13.3) | 325 (27.1) | 1170 (13.3) | 2340 (16.5)

4. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to 168h Postdose (AUC0-168h) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5 and 8
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
hr.µg/mL | 78.0 (22.5) | 350 (14.2) | 807 (28.5) | 2940 (11.6) | 6190 (13.1)

5. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Zero to the Last Measurable Concentration (AUC0-last) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
hr.µg/mL | 86.9 (21.9) | 402 (14.4) | 933 (30.7) | 3380 (11.5) | 7070 (10.9)

6. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve Extrapolated to Infinity (AUC0-inf)
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr.µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
hr.µg/mL | 89.1 (21.7) | 417 (13.7) | 947 (29.3) | 3380 (11.5) | 7080 (10.9)

7. Secondary Outcome: Terminal Rate Constant (Lambda z) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: (1/h)
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
(1/h) | 0.0103 (19.7) | 0.00625 (57.0) | 0.00690 (59.0) | 0.00409 (19.5) | 0.00436 (21.8)

8. Secondary Outcome: Apparent Terminal Half-Life (T1/2) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
hr | 67.1 (19.7) | 111 (57.0) | 100 (59.0) | 170 (19.5) | 159 (21.8)

9. Secondary Outcome: Total Body Clearance Calculated as Dose/AUC (CL) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/hr/kg
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
mL/hr/kg | 1.14 (21.3) | 0.965 (13.8) | 1.28 (29.4) | 1.07 (10.9) | 1.03 (11.1)

10. Secondary Outcome: Volume of Distribution at Steady-State (Vss) of RO7126209
Description: as for outcome 3
Time Frame: Days 1, 2, 3, 4, 5, 8, 10, 15, 22, 29, 43 and 57
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/kg
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 5
mL/kg | 88.6 (25.1) | 90.3 (26.3) | 108 (35.5) | 88.7 (22.6) | 85.3 (22.8)

11. Secondary Outcome: Cerebrospinal Fluid (CSF) Concentration of RO7126209
Description: RO7126209 CSF concentrations were measured by a specific and validated method. Geometric Mean and Coefficient of Variation data are presented below.
Time Frame: Day 3 and Day 5
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3
µg/mL
  Day 3 | 0.00414 (33.0) | 0.0202 (26.5) | 0.047 (29.4) | 0.105 (40.3) | 0.284 (35.9)
  Day 5: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2
  Day 5 | 0.00228 (18.7) | 0.0126 (26.1) | 0.0274 (22.9) | 0.0755 (7.4) | 0.151 (9.8)

12. Secondary Outcome: Percentage of Participants With Anti-RO7126209 Antibodies (ADAs)
Description: The numbers and proportions of Anti-Drug Antibody (ADA) positive participants and ADA negative participants at baseline (baseline prevalence) and after study drug administration (post-baseline incidence during both the treatment and follow-up periods) were summarized per dose group during both the treatment and follow-up period.
Time Frame: Days 1, 8, 29 and 57
Population: The Immunogenicity population was defined as all participants who had at least one pre-dose or at least one post dose ADA assessment and were included and analysed according to the treatment they actually received. Data presented below is only for participants included in the actual analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
Number analyzed (Participants) | 4 | 4 | 6 | 6 | 6
Percentage of Participants | 50.0 | 25.0 | 66.7 | 83.3 | 83.3

ADVERSE EVENTS:
Time Frame: Up to approximately 9 weeks
Arm/Group | Placebo | RO7126209 (0.1 mg/kg) | RO7126209 (0.4 mg/kg) | RO7126209 (1.2 mg/kg) | RO7126209 (3.6 mg/kg) | RO7126209 (7.2 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 8/10 | 3/4 | 2/4 | 5/6 | 6/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | RO7126209 (0.1 mg/kg) (N=4) | RO7126209 (0.4 mg/kg) (N=4) | RO7126209 (1.2 mg/kg) (N=6) | RO7126209 (3.6 mg/kg) (N=6) | RO7126209 (7.2 mg/kg) (N=6)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Crepitations (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (4) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 0 (0) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/94/NCT04023994/Prot_SAP_000.pdf